CLINICAL TRIAL: NCT01351012
Title: Canola and Flax Oils in Modulation of Vascular Function and Biomarkers of Cardiovascular Disease Risk
Brief Title: Canola Oil Multicentre Intervention Trial
Acronym: COMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Toronto (Other); Penn State University (Other); Laval University (Other)
Responsible Party: Principal Investigator, Dr. Peter Jones, Director of the Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2010:047
Record Dates: First submitted 2011-03-14; First posted 2011-05-10 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Metabolic Syndrome
Keywords: Canola oil; High oleic canola oil; Flax oil; ALA; DHA; Metabolic syndrome; Cardiovascular disease; Endothelial function; FADS1; Gut microbiome; Body composition; Psychosocial status; Cholesterol; Lipids; Lipoproteins; Inflammation; Lipid peroxidation
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Inflammation | interventions — Safflower Oil; Rapeseed Oil; Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Corn and safflower oil (Placebo Comparator)
  Interventions: Other: Corn and safflower oil
- Canola oil (Active Comparator)
  Interventions: Other: Canola oil
- High oleic acid canola oil (Active Comparator)
  Interventions: Other: High oleic acid canola oil
- DHA enriched high oleic acid canola oil (Active Comparator)
  Interventions: Other: DHA enriched high oleic acid canola oil
- Flax and safflower oil (Active Comparator)
  Interventions: Other: Flax and safflower oil

INTERVENTIONS:
Other: Corn and safflower oil — The oil (60 g/d/3000 kcal) is given in two daily fruit shakes for 4 weeks
  Arms: Corn and safflower oil
Other: Canola oil — The oil (60 g/d/3000 kcal providing 3.8 g ALA) is given in two daily fruit shakes for 4 weeks
  Arms: Canola oil
Other: High oleic acid canola oil — The oil (60 g/d/3000 kcal providing 41.2 g oleic acid and 1.2 g ALA) is given in two daily fruit shakes for 4 weeks
  Arms: High oleic acid canola oil
Other: DHA enriched high oleic acid canola oil — The oil (60 g/d/3000 kcal providing 1.2 g of ALA and 3.6 g of DHA) is given in two daily fruit shakes for 4 weeks
  Arms: DHA enriched high oleic acid canola oil
Other: Flax and safflower oil — The oil (60 g/d/3000 kcal providing 6.9 g of ALA) is given in two daily fruit shakes for 4 weeks
  Arms: Flax and safflower oil

SUMMARY:
The purpose of the study is to examine how the consumption of different dietary oil varieties affects a broad range of metabolic responses that are important in the development of cardiovascular diseases. This study will examine the relationship between dietary oil consumption and arterial function, blood fat content, and blood markers of cardiovascular disease risk. Additionally, the efficiency of the body in converting fat from dietary oils into other specific fat compounds with know health benefits will be examined. Also, the correlation between psychosocial parameters and vascular function will be studied.

DETAILED DESCRIPTION:
Although consumption of omega-3 fatty acids favorably modulate circulating lipids and arterial health, there is confusion surrounding the specific health benefits of plant based alpha-linolenic acid (ALA) versus marine derived eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). This research will examine the health benefits of ALA from consumption of diets rich in canola oil, novel monounsaturated fatty acid (MUFA) and DHA enriched canola oils, and flax oil compared with a control diet representative of North American diets rich in omega-6 and saturated fats. Treatment oils will be examined for potential influence on endothelial dysfunction, inflammation, oxidation, body composition, and plasma lipoprotein characterization. Furthermore, in an effort to elucidate the genetic factors that promote ALA conversion to EPA/DHA and strengthen the role of ALA in cardiovascular health, a major objective is to correlate common genetic variants in the fatty acid desaturase 1 (FADS1) and fatty acid desaturase 2 (FADS2) gene cluster with ALA conversion to EPA/DHA and n-3 fatty acid composition of serum phospholipids in response to consumption of the treatment oils. Besides, psychosocial predictors of vascular function will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥94 cm (males) or ≥80 cm (females)

plus at least one of the following:

* Triglycerides ≥1.7 mmol/L
* High density lipoprotein (HDL) cholesterol <1 mmol/L (males) or <1.3 mmol/L (females)
* Low density lipoprotein (LDL) cholesterol ≥3.5 mmol/L
* Blood pressure ≥130 mmHg (systolic) and/or ≥85 mmHg (diastolic)
* Glucose ≥5.5 mmol/L

Exclusion Criteria:

* Thyroid disease
* Diabetes mellitus
* Kidney disease
* Liver disease
* Smoking
* Heavy drinking
* Use of medication known to affect lipid metabolism during the last 3 months(cholestyramine, colestipol, niacin, clofibrate, gemfibrozil, probucol, HMG CoA reductase inhibitors)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | Endothelial function will be measured at baseline and at the end of each of the five 4-week treatment phases over a period of nine months.
  Non-invasive peripheral arterial tonometry (EndoPAT) is used to assess endothelial function.

SECONDARY OUTCOMES:
Change in ALA conversion to EPA/DHA | Blood samples will be collected at the end of each of the five 4-week treatment phases over a period of nine months.
  On day 28 of each experimental phase, a fasting baseline blood sample is taken prior to administration of an oral dose of deuterium oxide containing a higher than normal proportion of the hydrogen isotope deuterium (2H). Fasting blood samples will be obtained 24 h following the tracer dose. Enrichment of 2H in EPA and DHA plasma triglycerides, non-esterified fatty acids, and phosphatidylcholine will be measured by GC-combustion isotope-ratio mass spectrometry.
Change in body composition | Measurements will be done at the start and end of each of the five 4-week treatment phases over a period of nine months.
  Changes in body composition will be assessed using dual-energy X-ray absorptiometry (DXA) scans. Also, a MRI scan will be performed on each subject at the start of the study.
Change in FADS 1 & 2 mRNA and protein expression | Blood samples will be collected at the end of each of the five 4-week treatment phases over a nine-month period.
  mRNA and protein expression of genes/proteins involved in fatty acid metabolism will be analyzed using standard RT-PCR and immunoblotting protocols.
Change in psychosocial correlates | Measurements are done at baseline, at the start of the fifth treatment phase and at the end of each of the five 4-week treatment phases.
  Subjects will complete questionnaires regarding their mood and recent sleep (state questionnaires) and a questionnaire regarding their overall mood, social support and behaviors (trait questionnaire).
Change in plasma lipids and lipoproteins, inflammatory cytokines and peroxidation biomarkers | Blood samples are collected at the start and end of each of the five 4-week treatment phases over a nine-month period.
Blood Pressure | Over 3 years; at baseline and endpoint of each 4-week treatment phases
  Blood pressure data (change in both systolic and diastolic) was taken 3 times at the baseline and endpoint of each phase of the trial. 2nd and 3rd measures were averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Study Chair — University of Manitoba; David Jenkins, PhD, Principal Investigator — University of Toronto; Penny Kris-Etherton, PhD, RD, Principal Investigator — Penn State University; Sheila West, PhD, Principal Investigator — Penn State University; Benoit Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Liu X, Garban J, Jones PJ, Vanden Heuvel J, Lamarche B, Jenkins DJ, Connelly PW, Couture P, Pu S, Fleming JA, West SG, Kris-Etherton PM. Diets Low in Saturated Fat with Different Unsaturated Fatty Acid Profiles Similarly Increase Serum-Mediated Cholesterol Efflux from THP-1 Macrophages in a Population with or at Risk for Metabolic Syndrome: The Canola Oil Multicenter Intervention Trial. J Nutr. 2018 May 1;148(5):721-728. doi: 10.1093/jn/nxy040. PMID 30053283
- [Derived] Liu X, Kris-Etherton PM, West SG, Lamarche B, Jenkins DJ, Fleming JA, McCrea CE, Pu S, Couture P, Connelly PW, Jones PJ. Effects of canola and high-oleic-acid canola oils on abdominal fat mass in individuals with central obesity. Obesity (Silver Spring). 2016 Nov;24(11):2261-2268. doi: 10.1002/oby.21584. PMID 27804268
- [Derived] Jones PJ, MacKay DS, Senanayake VK, Pu S, Jenkins DJ, Connelly PW, Lamarche B, Couture P, Kris-Etherton PM, West SG, Liu X, Fleming JA, Hantgan RR, Rudel LL. High-oleic canola oil consumption enriches LDL particle cholesteryl oleate content and reduces LDL proteoglycan binding in humans. Atherosclerosis. 2015 Feb;238(2):231-8. doi: 10.1016/j.atherosclerosis.2014.12.010. Epub 2014 Dec 9. PMID 25528432
- [Derived] Baril-Gravel L, Labonte ME, Couture P, Vohl MC, Charest A, Guay V, Jenkins DA, Connelly PW, West S, Kris-Etherton PM, Jones PJ, Fleming JA, Lamarche B. Docosahexaenoic acid-enriched canola oil increases adiponectin concentrations: a randomized crossover controlled intervention trial. Nutr Metab Cardiovasc Dis. 2015 Jan;25(1):52-9. doi: 10.1016/j.numecd.2014.08.003. Epub 2014 Aug 20. PMID 25240692
- [Derived] Jones PJ, Senanayake VK, Pu S, Jenkins DJ, Connelly PW, Lamarche B, Couture P, Charest A, Baril-Gravel L, West SG, Liu X, Fleming JA, McCrea CE, Kris-Etherton PM. DHA-enriched high-oleic acid canola oil improves lipid profile and lowers predicted cardiovascular disease risk in the canola oil multicenter randomized controlled trial. Am J Clin Nutr. 2014 Jul;100(1):88-97. doi: 10.3945/ajcn.113.081133. Epub 2014 May 14. PMID 24829493
- [Derived] Senanayake VK, Pu S, Jenkins DA, Lamarche B, Kris-Etherton PM, West SG, Fleming JA, Liu X, McCrea CE, Jones PJ. Plasma fatty acid changes following consumption of dietary oils containing n-3, n-6, and n-9 fatty acids at different proportions: preliminary findings of the Canola Oil Multicenter Intervention Trial (COMIT). Trials. 2014 Apr 23;15:136. doi: 10.1186/1745-6215-15-136. PMID 24754911